CLINICAL TRIAL: NCT01880190
Title: Volume Replacement With HES 130/0.4 Attenuates Inflammatory Response to Major Abdominal Surgery Compared to Ringer's Lactate (RL); the Effect on Cytokines and Matrix Metalloproteinases
Brief Title: A Comparative Study of Volume Replacement With HES 130/0.4 Versus Ringer's Lactate (RL) Regarding Their Effects on Inflammatory Biomarkers (Cytokines and Matrix Metalloproteinases) Responses to Major Abdominal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paraskevi Matsota (Other)
Responsible Party: Sponsor-Investigator, Paraskevi Matsota, Assistant Professor of Anesthesiology, MD, PhD, Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 301
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Inflammation
MeSH Terms: interventions — Ringer's Lactate; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Ringer's Lactate (Active Comparator): Crystalloid solution
  Interventions: Other: Ringer's Lactate
- HES 130/0.4 and Ringer's Lactate (Active Comparator): Colloid solution
  Interventions: Other: HES 130/0.4 and Ringer's Lactate

INTERVENTIONS:
Other: Ringer's Lactate
  Arms: Ringer's Lactate
Other: HES 130/0.4 and Ringer's Lactate
  Arms: HES 130/0.4 and Ringer's Lactate

SUMMARY:
Various stimuli such as trauma, infection and major surgery may alter the physiologic immune balance and initiate systemic inflammatory processes. This pathophysiological event is characterized by the release of potent inflammatory mediators into the circulation.

Among these, pro- and anti-inflammatory cytokines such as interleukin-6 (IL-6), IL-8 or IL-10, ICAM-1 play a dominant role as local or systemic regulators in the acute inflammatory response. Recent studies have also investigated the role of matrix metalloproteinases (MMPs) in the inflammatory response. The MMPs constitute a family of enzymes that are structurally related neutral proteinases. MMPs can degrade essentially all extracellular matrix (ECM) components and play an important role in wound healing and remodeling of the ECM. The Tissutal Inhibitor MetalloProteine (TIMPs) are important regulator of MMPs activity.

The inflammatory response coming of surgery mainly affects surgical patients' outcome. Many factors may attributed to this response, such as the kind of operation, the extent of surgical trauma, the patient's medical history and therapy, as well as the type of anesthesia used. Apart from that, the kind of fluids administered for volume replacement was revealed to alter the inflammatory processes. Several studies have addressed on this issue mainly involved abdominal surgery and provided compelling evidence that perioperative fluid optimization produces benefits for the patient, with regard to inflammatory biomarkers such as cytokines, matrix metalloproteinases, intercellular adhesion molecule-1(ICAM-1). They support that the different volume replacement strategies, using only crystalloids or combination of crystalloids with colloids (HES 130/0,4), may have important impact on immune response. However, the relevant studies investigated different inflammatory biomarkers, and usually involved either metalloproteinases, and their inhibitors (TIMPs) or cytokines.

In our study we investigated the hypothesis that intra- and postoperative volume replacement with HES attenuates inflammatory response to elective abdominal surgery compared to RL fluid therapy. For this purpose both metalloproteinases, MMP-9, MMP-13, their inhibitor, TIMP-1, cytokines, IL-6, IL-8 and the intercellular adhesion molecule-1, ICAM-1 were investigated postoperatively. Their changes during the first 24 postoperative hours consisted our primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I and ASA II

Exclusion Criteria:

* cardiac insufficiency ( > New York Heart Association (NYHA) class II)
* renal insufficiency (serum creatinine > 200μm/L)
* severe pulmonary disease (chronic obstructive lung disease, PaO2 < 70 mmHg when FiO2= 0.21)
* liver disfunction (AST > 40 U/L, ALT > 40 U/L)
* diabetes mellitus
* autoimmune disease
* pre-existing signs of bacterial (WBC > 10000, body temperature > 38.0 C)or viral infection (HBV, HCV, HIV, CMV)
* pre-existing signs of active inflammation (CRP > 4)
* malignant neoplasia
* morbid obesity
* patients in extreme muscular activity (athletes)
* patients with chronic use of corticosteroids or β- blockers or non-steroid anti-inflammatory substances
* known allergic reactions to colloids solutions

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Measurement of inflammatory biomarkers (MMP-9, MMP-13, TIMP-1, IL-6, IL-8 ICAM-1) in abdominal surgery. | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece